CLINICAL TRIAL: NCT00669292
Title: Phase I/II Study of URLC10-177 and TTK-567, Novel Tumor Specific Epitope Peptides Restricted to HLA-A*2402 Derived From Tumor Associated Antigens, Combined With CpG7909, a TLR9 Agonist, in Patients With Advanced or Recurrent Esophageal Cancer.
Brief Title: PhaseⅠ/Ⅱ Study of URLC10-177 and TTK-567 Peptide Vaccine Combined With CpG7909 in Patients With Esophageal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wakayama Medical University (Other)
Collaborators: Human Genome Center, Institute of Medical Science, University of Tokyo (Other)
Responsible Party: Second Department of Surgery, Wakayama Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WEUTC
Record Dates: First submitted 2008-04-28; First posted 2008-04-30 (Estimated); Last update posted 2010-09-09 (Estimated); Status verified 2010-09

CONDITIONS: Esophageal Cancer
Keywords: esophageal cancer; peptide; URLC10; TTK; CpG7909
MeSH Terms: conditions — Esophageal Neoplasms | interventions — ProMune

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: URLC10-177, TTK-567, CpG-7909 — peptide, peptide, TLR-9 agonist

SUMMARY:
This is a single institution phase I / II trial to evaluate the safety and efficacy of URLC10-177 and TTK-567 emulsified with Montanide ISA 51 in combination with different doses of CpG7909 in patients with advanced or recurrent esophageal cancer.

DETAILED DESCRIPTION:
phase I: Patients will be vaccinated on day 1,8,15 and 22 of each 28-day treatment cycles. On each vaccination day, the URLC10-117 peptide(1mg) and TTK-567 peptide(1mg) mixed with CpG 7909 (escalating doses: 0, 0.02, 0.1mg/kg) emulsified with Montanide ISA 51 will be administered by subcutaneous injection. Repeated cycles of vaccine will be administered until patients develop progressive disease or unacceptable toxicity, or for maximum 2 cycles, whichever occurs first. In this phase I study, we evaluate the safety and tolerability of URLC10-177, TTK-567 and different doses of CpG7909 to determine the recommended phase II dose of CpG7909.

phase II: Patients will be vaccinated on day 1,8,15 and 22 of each 28-day treatment cycles. On each vaccination day, the URLC10-117 peptide(1mg) and TTK-567 peptide(1mg) mixed with CpG 7909 (recommended dose determined in phase I study) emulsified with Montanide ISA 51 will be administered by subcutaneous injection. Repeated cycles of vaccine will be administered for 2 cycles. In this phase II study, we evaluate the efficacy of this vaccine therapy.

ELIGIBILITY:
Inclusion Criteria:

DISEASE CHARACTERISTICS

1. locally advanced or metastatic esophageal cancer precluding curative surgical resection and recurrent esophageal cancer
2. measurable disease by CT scan

PATIENT CHARACTERISTICS

1. ECOG performance status 0-1
2. Life expectancy > 3 months
3. Laboratory values as follows

   * 2000/mm3 < WBC < 15000/mm3
   * Platelet count > 75000/mm3
   * Aspartate transaminase < 150 IU/L
   * Alanine transaminase < 150 IU/L
   * Creatinine < 2.0 mg/dl
4. HLA-A*2402
5. Able and willing to give valid written informed consent

Exclusion Criteria:

1. Pregnancy(woman of childbearing potential:Refusal or inability to use effective means of contraception)
2. Breastfeeding
3. Active or uncontrolled infection
4. Concurrent treatment with steroids or immunosuppressing agent
5. Prior chemotherapy,radiation therapy, or immunotherapy within 4 weeks
6. Clinically significant heart disease
7. Decision of unsuitableness by principal investigator or physician-in-charge

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2006-11; Primary Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Safety(Phase I:toxicities as assessed by NCI CTCAE version3) and efficacy(Phase II:Feasibility as evaluated by RECIST) | 2 months

SECONDARY OUTCOMES:
To evaluate immunological responses (Phase I/II) | 2months
To determine the recommended phase II dose of CpG7909(Phase I) | 2months
To determine the clinical effectiveness in the patients with measurable disease(Phase I) | 2months
To analyze the toxicity(Phase II) | 2months
Time to progression(Phase II) | 5 years
survival(Phase II) | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Wakayama Medical University Hospital, 811-1 Kimiidera, Wakayama, Wakayama, Japan

REFERENCES:
- [Derived] Iwahashi M, Katsuda M, Nakamori M, Nakamura M, Naka T, Ojima T, Iida T, Yamaue H. Vaccination with peptides derived from cancer-testis antigens in combination with CpG-7909 elicits strong specific CD8+ T cell response in patients with metastatic esophageal squamous cell carcinoma. Cancer Sci. 2010 Dec;101(12):2510-7. doi: 10.1111/j.1349-7006.2010.01732.x. Epub 2010 Sep 28. PMID 20874827